CLINICAL TRIAL: NCT04249557
Title: Exercise is Medicine: a Cohort Study
Acronym: EIM-cohort
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Lee Kam Pui, Clinical Assistant Professor, Chinese University of Hong Kong
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EIM-cohort
Record Dates: First submitted 2020-01-21; First posted 2020-01-31 (Actual); Last update posted 2024-07-16 (Actual); Status verified 2024-07

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- EIM group (Experimental): This contains: A 12-week Exercise is medicine teaching class containing 6-18 patients per group (class size may be limited by social distancing policy in Hong Kong), homework are prescribed to participants to encourage regular exercise. The exercise level will be recorded by a tracker and provides feedback to the participants and physical trainer. The physical parameters such as fat percentage and blood pressure level will be feedback to the patients to encourage exercise. (If sports center are closed by the Government, the classes will be conducted online)
  Interventions: Behavioral: exercise is medicine

INTERVENTIONS:
Behavioral: exercise is medicine — a 12-week exercise classes program combined with other motivational skills, including feedback and information technology support. The whole program lasts for 1 year for each participant

SUMMARY:
6,000 patients with HT and/or DM will be recruited to participate a 12-week EIM exercise intervention, which also involve consistent feedback and reminders using information technology (IT). The primary outcome will be improvement of blood pressure at 1-year. Other clinical outcomes will be obtained on recruitment (baseline), 12-week (immediately after EIM classes) and 1-year after recruitment

ELIGIBILITY:
Inclusion Criteria:

* have a clinical diagnosis of primary HT and/or type II DM from clinical medical record
* having less than 150 minutes of moderate intensity exercise per week OR having less than 75 minutes of intensive intensity exercise per week (this is set according to latest World Health Organization guideline)
* who have used any mobile apps on their phone (because the intervention involve use of apps to monitor and remind regular exercise)

Exclusion Criteria:

* patients with diagnosed chronic obstructive lung disease and recent stroke (within last 12 months)
* Patients on 3 or more anti-hypertensive medications (on maximum or maximal tolerable doses) are excluded because these patients have resistant HT and may represent another spectrum of disease.
* Patients with spinal cord compression, radiculopathy with active pain, or osteoarthritis of hips and knees that are on the waiting list for joint replacement surgery are excluded for safety reasons.
* acute myocardial infarction in last 6 months
* ongoing angina
* uncontrolled cardiac arrhythmia
* acute diseases including known active endocarditis/acute pulmonary embolism, pulmonary infarction, deep vein thrombosis, acute aortic dissection, acute myocarditis
* known aortic stenosis
* known heart failure
* known obstructive left main coronary artery stenosis
* uncontrolled ventricular rates
* complete heart block
* known hypertrophic obstructive cardiomyopathy
* mental impairment that limit co-operation
* resting blood pressure with systolic blood pressure >180mmHg or diastolic blood pressure >110mmHg
* known anaemia with haemoglobin level less than 11gm/dL
* known uncorrected electrolyte imbalance
* known uncontrolled hyperthyroidism.
* For DM patients, patients with proliferative diabetic retinopathy and recent retinal bleeding (in last 12 months)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6000 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2024-05-30 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
office blood pressure | Change from Baseline Systolic Blood Pressure at 3 months
  office systolic blood pressure

SECONDARY OUTCOMES:
serum lipid level | baseline, 3-month after recruitment (immediate after EIM class), 12-month after recruitment (end-of-study)
  low density lipoprotein, high density lipoprotein, total cholesterol, triglyceride
body fat percentage | baseline, 3-month after recruitment (immediate after EIM class), 12-month after recruitment (end-of-study)
  that will be measured by a validated machine
body mass index | baseline, 3-month after recruitment (immediate after EIM class), 12-month after recruitment (end-of-study)
  body weight (in kilogram) divided by square of body height (in meter)
international physical activity questionnaire- short form | baseline, 3-month after recruitment (immediate after EIM class), 12-month after recruitment (end-of-study)
  assess the amount of exercise, physical activities and sitting time in the last 7 days. After asking the number of hours spent on walking, moderate intensity exercise and vigorous exercise, the amount of energy expenditure (in the unit MET-min/week) can be calculated. The higher the number, the higher the energy expenditure
office blood pressure | baseline, 12-month after recruitment (end-of-study)
  office systolic and diastolic blood pressure

CONTACTS AND LOCATIONS:
Locations (1):
- Lek Yuen Clinic, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided
Can share out after personal permission is obtained